CLINICAL TRIAL: NCT06784362
Title: Diagnostic and Prognostic Test for Periodontitis and Peri-implantitis (AHC-FRDgrant)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: #1511M79922
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Periodontal Diseases; Periodontitis; Peri-Implantitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gingival fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy group: individuals without periodontitis or peri-implantitis
  Interventions: Other: No intervention
- untreated group: individuals with periodontitis or peri- implantitis who have been informed of the need for treatment - but have decided not to have treatment (untreated group)
  Interventions: Other: No intervention
- high risk group: individuals who received treatment for periodontitis or peri-implantitis and are now receiving regular dental hygiene care every 3 months (high risk group).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
The dental community, dental insurance companies and the public are becoming increasingly aware of the high prevalence of gum disease around teeth (periodontitis) and around dental implants (peri-implantitis). To date, it cannot be accurately predicted which individuals will develop or re-develop periodontitis or peri-implantitis, leading most dental patients to undergo unnecessary treatment and undue risks and costs. Gingival fluid is a serum-like fluid that diffuses into the oral cavity by flowing between the gum and the tooth or dental implant.

Oral bacteria that grow around teeth and dental implants induce inflammation and change the amount and composition of the gingival fluid. The study hypothesizes that the spectra of metabolites in the inflammatory transudates and exudates around teeth and dental-implants are predictors of future periodontitis or peri-implantitis. The first objective is to use proton nuclear magnetic resonance (H-NMR) spectroscopy in a cross-sectional study to map mapping the metabolites in the gingival fluid that are capable of discriminating between healthy gum tissue and gum tissue that shows signs of periodontitis or dental peri-implantitis. The second objective is to begin prospective measurement of gingival fluid metabolites every 6 months in (i) individuals without periodontitis or peri-implantitis (healthy group), (ii) individuals with periodontitis or peri- implantitis who have been informed of the need for treatment - but have decided not to have treatment (untreated group) and (iii) individuals who received treatment for periodontitis or peri-implantitis and are now receiving regular dental hygiene care every 3 months (high risk group). By defining metabolites that can discriminate health from disease (Aim 1) and by measuring proportional changes of key metabolites relative to disease progression over time (Aim 2), the study will be able to predict in a site-specific manner, (a) the risk of disease initiation in people who do not initially have periodontitis or peri-implantitis (healthy persons), and (b) disease progression in untreated people or in people who were treated and are currently in a dental hygiene maintenance program. Accomplishing these two aims will provide a foundation from which to increase the efficacy of prevention whilst abating the morbidity and cost associated with current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with disease (cases) were diagnosed with generalized chronic severe periodontitis with at least five teeth having clinical evidence of disease [clinical attachment loss (CAL) ≥ 5mm, at least one site with probing depth (PD) ≥ 7 mm] and radiographic evidence of at least 30% bone loss
* Control subjects exhibited a healthy periodontium (no PD >3 mm. no site with CAL) with no radiographic evidence of bone loss.
* Case and control subjects were in good general health.

Exclusion Criteria:

* uncontrolled systemic disease, such as diabetes;
* systemic antibiotic use within the past 3 months;
* unable to provide consent; and
* history of periodontal treatment or local antibiotic use in the past 12 months;
* use of NSAIDs in the past 3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with disease (cases) were diagnosed with generalized chronic severe periodontitis with at least five teeth having clinical evidence of disease [clinical attachment loss (CAL) ≥ 5mm and at least one site with probing depth (PD) ≥ 7 mm], and radiographic evidence of at least 30% bone loss. Control subjects exhibited a healthy periodontium (no PD >3 mm. no site with CAL) with no radiographic evidence of bone loss. Case and control subjects were in good general health. Smoking habits were noted. Case and control exclusion criteria included: 1) uncontrolled systemic disease, such as diabetes; 2) systemic antibiotic use within the past 3 months; 3) unable to provide consent; and 4) history of periodontal treatment or local antibiotic use in the past 12 months; 5) use of NSAIDs in the past 3 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
defining metabolites that can discriminate health from disease | 6, 12, 18, 24 months
  Gingival fluid samples using use proton nuclear magnetic resonance (H-NMR) spectroscopy, every 6 months for 24 months
measuring proportional changes of key metabolites relative to disease progression over time | 6, 12, 18, 24 months
  Gingival fluid samples using use proton nuclear magnetic resonance (H-NMR) spectroscopy, every 6 months for 24 months